CLINICAL TRIAL: NCT04830150
Title: The Effect of Supportive Nursing Interventions on Reducing Stress Levels of Mothers of Infants in Neonatal Intensive Care Unit: A Randomized Controlled Trial
Brief Title: The Effect of Supportive Nursing Interventions of Mothers of Infants in Neonatal Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Dilekkucu Kalemdar, PhD, RN, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 95531838-663.05
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Stress, Psychological
Keywords: cortisol; mother; neonatal intensive care; neonate; stress; supportive intervention
MeSH Terms: conditions — Stress, Psychological | interventions — Intensive Care Units, Neonatal

STUDY DESIGN:
Intervention Model Description: This study was a prospective, pre-and post-test randomised controlled trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supportive interventions group (Experimental): Supportive and educational nursing interventions about reducing maternal stress levels in the experimental group included the following: the NICU was physically described to mothers on the first day they visited their infants, mothers were introduced to team members, and given information about how to obtain information about their baby, visiting hours and conditions.
  Interventions: Behavioral: Supportive interventions on the stress levels of mothers of infants hospitalized in the Neonatal Intensive Care Unit (NICU).
- control group (No Intervention): Mothers did not have any other intervention applied by the researchers during routine operation while their infants were in the unit.

INTERVENTIONS:
Behavioral: Supportive interventions on the stress levels of mothers of infants hospitalized in the Neonatal Intensive Care Unit (NICU). — This study was conducted to determine the effects of supportive interventions on the stress levels of mothers of infants hospitalized in the Neonatal Intensive Care Unit (NICU).
  Arms: supportive interventions group

SUMMARY:
Objective: This study was conducted to determine the effects of supportive interventions on the stress levels of mothers of infants hospitalized in the Neonatal Intensive Care Unit (NICU).

Backround: The inability to nurture the healthy baby dreamed of, disease and intensive care processes are situations causing a crisis for parents. The stress experienced by mothers may affect emotional status and the foundation of the mother-ınfant attachment. For this reason, mothers of infants hospitalized in the NICU need support to cope with the stressful events they experience.

Design: This study was a prospective, pre-and post-test randomised controlled trial. Methods: The population of the research comprised mothers with neonates admitted to the NICU of a state hospital, abiding by the sample selection criteria and who accepted participation in the research. The research was completed with 85 mothers in two groups of 45 subjects and 40 controls selected at random. Data collection used the Parental Stressor Scale: Neonatal Intensive Care Unit (PSS:NICU), NICU Parent Belief Scale (NICU:PBS), State-Trait Anxiety Inventory (STAI TX-2) and saliva cortisol analysis.

DETAILED DESCRIPTION:
This study was performed with the aim of determining the effect of supportive interventions on maternal stress levels among mothers with infants hospitalized in the NICU.

This was a randomized pre- and post-test controlled trial was conducted to determined the effect of planned educational and supportive nursing interventions given to mothers with infants in the NICU on the stress, anxiety and beliefs of mothers in the NICU of Women and Pediatrics Training and Research Hospital. This study was conducted at a state hospital's NICU in the east part of Turkey. According to the criteria of the T.R. Ministry of Health, the unit in which the study was performed was a Level I NICU. The unit had 10 incubators and 10 nurses were employed in the NICU. The nurses in the NICU worked in groups of three, in two shifts, providing care and treatment of the newborns in the unit. This part of Turkey is geographically located in a rural area in the east. The mothers with infants in the NICU were informed by the physicians and nurses on certain days of the week about the hours at which they were allowed to visit their infants.

Power analysis of the sample number used the G*Power (v. 3.1.9.2) program and was based on previous studies. According to Jacob Cohen's effect size coefficients, assuming large effect size in assessments between two independent groups (d=0.40), with α=0.05 and 1-β=0.95 (90% power), each group was required to contain at least 39 people. Considering data loss, each group included 50 mothers. As saliva samples were insufficient in 10 mothers in the experiment group and 5 mothers in the control group, this data was excluded from the study. The research was completed with 85 mothers, comprising 40 subjects and 45 controls chosen at random (Fig. 1).

2.3. Randomization: sequence generation, type, allocation concealment mechanism, and implementation Randomization was performed using a computer program. The participants were randomised and assigned by a researcher into two groups using the Integer Generator free software (www.random.org), which produces random numbers in configurable intervals: 40 in intervention group and 45 in control group.

Data collection used the "Mother and Neonate Descriptive Information Form", "Parental Stressor Scale: Neonatal Intensive Care Unit (PSS:NICU)", "NICU Parent Belief Scale (NICU PBS)", State-Trait Anxiety Inventory (STAI TX-2)" and "saliva cortisol analysis".

Before the mothers first visits to their infants, the mother and neonate descriptive information form, PSS: NICU, STAI TX-2 and NICU Parent Belief scale were completed by the researcher during face-to-face interviews with the mother and first saliva samples were taken from mothers. Mothers in the group with supportive nursing interventions completed the PSS:NICU, NICU-Parent Belief Scale and STAI-TX-2 again and had the post-test saliva sample taken when their infants were discharged from the NICU.

Supportive and educational nursing interventions about reducing maternal stress levels in the experimental group included the following: the NICU was physically described to mothers on the first day they visited their infants, mothers were introduced to team members, and given information about how to obtain information about their baby, visiting hours and conditions. Special tools and devices required for care like respiratory devices and monitors were described, and information was given about treatment of the neonate and general status. Mothers of neonates with appropriate clinical status were encouraged to touch their baby and hold their hand. Within the rules of the unit mothers were allowed to touch and hold their baby. Introduction to the NICU, informing about the baby and contact between mother and baby was completed within 30-45 minutes duration. As a guide to training, a 35-page "Care of your Baby in the Neonatal Intensive Care Unit" training booklet prepared by the researcher based on stress among families in the intensive care unit was given to mothers and included topics like the NICU environment, features of neonates born prematurely and at term, care, feeding, diseases, treatment methods, stress in the NICU, breastfeeding, preparation for discharge and baby care at home.

After the information session on the first visiting day for mothers and babies, seven interactive trainings were held each lasting nearly 90 minutes during the neonate's admission to hospital. During interactive training, power point presentations prepared by the researcher were presented on a large screen in the education salon in the hospital and arranged in two 45-minute sessions allowing mothers to share their experiences, excitement, sadness and worries. Planned nursing interventions were standardised for each mother with a check-list. Mothers were given information training about the NICU environment, features of babies born prematurely and at term, care, feeding, disease, treatment methods, stress in the NICU, breastfeeding, preparation for discharge and baby care at home. The relevant topics were chosen after relevant literature search by the researcher (Konukbay & Arslan, 2011; Lonio et al. 2016; Uludağ & Ünlüoğlu, 2012) and the second author's personal experience with parents of infants in the NICU. In the second session, the researchers gave training about positive thinking, healthy lifestyle, knowing yourself, stress management and relaxation techniques developed in the context of the literature within the scope of supportive nursing interventions for mothers (Nasiri et al., 2018; Nasiri et al., 2018). Mothers were taught the simple but powerful relaxation technique which is easy and can be performed nearly everywhere of deep breathing (diaphragmatic respiration). Each session began with this exercise and they were encouraged to perform it throughout the day.

During mothers first visits to their infants, mothers in this group had the mother and neonate descriptive information form, PSS: NICU, STAI TX-2 and NICU Parent Belief scale applied and first saliva samples were taken from mothers. Mothers did not have any other intervention applied by the researchers during routine operation while their infants were in the unit. When their infants were discharged from the NICU, mothers completed the PSS:NICU, NICU-Parent Belief Scale and STAI-TX-2 again and had the post-test saliva sample taken.

ELIGIBILITY:
Inclusion Criteria:

* Being aged between 20-40,
* having no chronic physical and psychological problems, being literate,
* no previously receiving training about the care of infants hospitalised in the NICU.

Exclusion Criteria:

* Having a gestational age of <28 and >37 weeks,
* Having a birth weight of 1500 grams less,

Ages: 28 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Parental Stressor Scale: Neonatal Intensive Care Unit (PSS:NICU) | Before the mothers first visits to their infants (the third day).
  This scale was developed by Miles, Funk and Carlson (1993) with the aim of determining the perceptions of parents about stressors due to the physical and psychosocial environment in the NICU. The scale uses a 5-point Likert score grading from 1 (not stressful) to 5 (excessively stressful).
Neonatal Infant Care Unit Parent Belief Scale (NICU PBS) | Before the mothers first visits to their infants (the third day).
  This scale developed by Melnyk et al. (2014) has three subdimensions (Parental Role Confidence, Parent-Baby Interaction, and Knowledge of the NICU) and includes a total of 18 items.
State-Trait Anxiety Scale (STAI TX-2) | Before the mothers first visits to their infants (the third day).
  The scale developed by Spielberger et al. in 1970 was adapted to Turkish with validity and reliability studies completed by Öner and Le Comte in 1983. The scale comprises 40 questions, with 20 questions about state and 20 questions about trait anxiety levels. In the research, 20 questions measuring trait anxiety were used. Expressions on the trait anxiety scale have choices of nearly never (1), sometimes (2), often (3), and nearly all the time (4). Items 21, 26, 27, 39, 33, 36 and 39 are inverse statements.
Saliva Cortisol Measurement | Before the mothers first visits to their infants (the third day).
  With the aim of determining cortisol levels in saliva, taking saliva samples with a kit is an easy and non-invasive method that does not cause stress (Kirschbaum & Hellhammer, 1994). Mothers were requested to avoid practices like eating-drinking and chewing gum for 30 minutes before the saliva collection procedure. Saliva samples were collected with special saliva test kits. Cotton from the kit is rotated within the mouth, cheeks and under the tongue for 1-2 minutes or chewed to complete the saliva collection procedure. Immediately after collecting saliva samples, they were centrifuged and stored at -20 degrees before transport to the laboratory. Saliva samples from mothers were taken from 08:00-10:00 in the morning.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Küçük Alemdar, Phd, Study Director — Ordu University
Locations (1):
- Dilek alemdar, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study was a prospective, pre-and post-test randomised controlled trial.

REFERENCES:
- [Derived] Yilmaz G, Kucuk Alemdar D. The Effect of Supportive Nursing Interventions on Reducing Stress Levels of Mothers of Infants in the Neonatal Intensive Care Unit: A Randomized Controlled Trial. Clin Nurs Res. 2022 Jun;31(5):941-951. doi: 10.1177/10547738211047359. Epub 2021 Sep 24. PMID 34555952